CLINICAL TRIAL: NCT05097209
Title: Camrelizumab Combined With Induction Chemotherapy and Intensity Modulated Radiotherapy for the Treatment of Locally Advanced Nasopharyngeal Carcinoma:a Randomized, Multicenter, Phase II Trial
Brief Title: Camrelizumab for the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Nanxishan Hospital (Unknown); Laibin People's Hospital (Other); Lingshan people's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Director, Department of Radiation Oncology, Principal Investigator, Clinical Professor, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-07
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Intensity Modulated Radiotherapy; Camrelizumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; spartalizumab; Gemcitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Camrelizumab 200mg will be given every 3 weeks for 3 cycles started on day 1 of induction chemotherapy and every 2 weeks for 9 cycles thereafter.
  Interventions: Drug: Camrelizumab; Drug: Gemcitabine; Drug: Induction Cisplatin; Radiation: intensity-modulated radiotherapy
- Chemoradiation arm (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT.
  Interventions: Drug: Gemcitabine; Drug: Induction Cisplatin; Radiation: intensity-modulated radiotherapy; Drug: Concurrent cisplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg will be given every 3 weeks for 3 cycles started on day 1 of induction chemotherapy and every 2 weeks for 9 cycles thereafter.
  Other Names: PD-1 antibody
  Arms: Camrelizumab arm
Drug: Gemcitabine — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation
  Other Names: Gem
Drug: Induction Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation
  Other Names: DDP
Radiation: intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
  Other Names: IMRT
Drug: Concurrent cisplatin — Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
  Other Names: DDP
  Arms: Chemoradiation arm

SUMMARY:
This trial plans to enroll patients with stage III-IVA (AJCC 8th, included T1-2N2-3 and/or T3-4N0-3 M0) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Patients will be randomized in a 1:1 ratio to receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation or 3 cycles of induction chemotherapy with gemcitabine and cisplatin and radiation plus Camrelizumab. All patients will receive intensity-modulated radiotherapy (IMRT). Camrelizumab will begin on day 1 of induction chemotherapy every 3 weeks for 3 cycles and continue every 2 weeks for 9 cycles.

DETAILED DESCRIPTION:
Objectives:To investigate the clinical efficacy of camrelizumab in the treatment of locoregionally-advanced nasopharyngeal carcinoma (LANPC).

Outline:Patients with stage III-IVA (AJCC 8th, included T1-2N2-3 and/or T3-4N0-3 M0) locoregionally-advanced nasopharyngeal carcinoma will be randomized in a 1:1 ratio to experimental arm and active comparator arm. Patients in experimental arm will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Camrelizumab 200mg will be given every 3 weeks for 3 cycles started on day 1 of induction chemotherapy and every 2 weeks for 9 cycles thereafter. Patients in active comparator arm will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed nasopharyngeal carcinoma.
2. Tumor staged as III-IVA (AJCC 8th, included T1-2N2-3 and/or T3-4N0-3 M0).
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥80g/L and platelet count ≥80×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Age > 70 or < 18.
2. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
3. Hepatitis C virus (HCV) antibody positive
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
6. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
7. Has a known history of interstitial lung disease.
8. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
9. Is pregnant or breastfeeding.
10. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
11. Has known allergy to large molecule protein products or any compound of camrelizumab.
12. Has a known history of human immunodeficiency virus (HIV) infection.
13. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  Calculated from randomization to the date of progression or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Calculated from randomization to the date of death from any cause.
Distant Metastasis-free survival (DMFS) | 3 years
  Calculated from randomization to the date of first distant metastasis.
Locoregional failure-free survival (LRRFS) | 3 years
  Calculated from randomization to the date of locoregional relapse.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, M.D., Principal Investigator — Wuzhou Red Cross Hospital; Yu-fei Pan, M.D., Principal Investigator — Guangxi Nanxishan Hospital; Yi-xin Su, M.D., Principal Investigator — Lingshan people's Hospital; Jian Zhang, M.D., Principal Investigator — Laibin People's Hospital
Locations (5):
- China (5):
  - Guangxi Nanxishan hospital, Guilin, Guangxi
  - Guilin Medical University, Guilin, Guangxi
  - Laibin People's Hospital, Laibin, Guangxi
  - Linshan people's hospital, Linshan, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

IPD SHARING:
Plan to Share IPD: No